CLINICAL TRIAL: NCT05266937
Title: A Phase II Trial of Atezolizumab Plus CArboplatin Plus Nab-paclitaxel as First-line Therapy in Metastatic Triple-negative PD-L1 Positive Breast Cancer Patients - the GIM25-CAPT Trial
Brief Title: Atezolizumab Plus CArboplatin Plus Nab-paclitaxel
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIM25-CAPT
Record Dates: First submitted 2020-02-10; First posted 2022-03-04 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Breast Cancer; Triple Negative Breast Cancer; PD-L1 Gene Mutation
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — atezolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: This is a Phase II, multicentre, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Single-arm study with the primary objective of providing preliminary evidence on the efficacy of atezolizumab plus carboplatin plus nab-paclitaxel as first-line therapy in metastatic triple-negative PD-L1 positive breast cancer patients as evaluated by % 2years OS.
  Interventions: Combination Product: Atezolizumab,Paclitaxel, Carboplatin

INTERVENTIONS:
Combination Product: Atezolizumab,Paclitaxel, Carboplatin — Atezolizumab at a fixed dose of 840 milligrams via intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle + Carboplatin area under the curve 2 via IV infusion on Days 1, 8, and 15 of each 28-day cycle + nab-Paclitaxel at a dose of 100 milligrams per square meter via IV infusion on Days 1, 8, and 15 of each 28-day cycle.
  In the absence of disease progression or unacceptable toxicity, study treatments will continue until the end of the study (2 years from last patient enrolled or study termination by the Sponsor).

SUMMARY:
Primary objective:

To provide preliminary evidence on the efficacy of atezolizumab plus carboplatin plus paclitaxel as first-line therapy in metastatic triple-negative PD-L1 positive breast cancer patients as evaluated by % 2years OS.

Secondary objective:

* To provide preliminary evidence on the efficacy of atezolizumab plus carboplatin plus paclitaxel as first-line therapy in metastatic triple-negative PD-L1 positive breast cancer patients in terms of % OS at 2.5 years
* To provide preliminary evidence on the efficacy of atezolizumab plus carboplatin plus paclitaxel as first-line therapy in metastatic triple-negative PD-L1 positive breast cancer patients in terms of % OS at 2 years in hormonal receptor (HR) between 1% and 10%
* To provide preliminary evidence on the efficacy of atezolizumab plus carboplatin plus paclitaxel as first-line therapy in metastatic triple-negative PD-L1 positive breast cancer patients in terms of post-progression survival
* To assess the activity of atezolizumab plus carboplatin plus paclitaxel as first-line therapy in metastatic triple-negative PD-L1 positive breast cancer patients in terms of ORR, and time to treatment failure
* To assess the safety of atezolizumab plus carboplatin plus paclitaxel as first-line therapy in metastatic triple-negative PD-L1 positive breast cancer patients

Exploratory Objectives:

Exploratory objectives will be focused on the assessment of both tumor-centered characteristics through the NGS analysis of circulating tumor DNA (ctDNA) and immune-centric features through the evaluation of a multiparametric Cancer agnostic circuLating ImmunOsignature (CLIO):

* To assess the association between patients' characteristics, treatment activity, efficacy and safety and through a CLIO in metastatic triple-negative breast cancer patients receiving atezolizumab plus carboplatin plus paclitaxel as first-line therapy
* To explore the association between the CLIO and treatment activity, efficacy and safety
* To explore the dynamics of circulating tumor DNA (ctDNA) levels and detectable aberrations with respect to treatment activity and efficacy Concomitant timepoints will not be used for cross-validations between the two methodologies.

DETAILED DESCRIPTION:
All eligible patients will receive carboplatin Area Under the Curve (AUC) 2 dd 1,8,15 q 28 dd, paclitaxel 90 mg/m2 dd 1,8,15 q 28 dd and atezolizumab 840 mg dd 1,15 q 28 dd and they will continue this treatment until progression of disease, unacceptable toxicity, death, withdrawal of consent, loss to follow-up, or study termination by the Sponsor. In case of interruption of one of the three drugs for unacceptable toxicity and/or medical decision, the patient may continue to receive one or more of the remaining drugs until progression per RECIST v1.1.

If the investigator decides to interrupt carboplatin and paclitaxel (for toxicity and/or medical decision), atezolizumab may be continued as maintenance therapy until disease progression or unacceptable toxicity.

All patients who discontinue study treatment (including due to PD) will be followed for survival approximately every 3 months for 2 years from last patient enrolled or until death, withdrawal of consent, loss to follow-up, or study termination by the Sponsor.

Imaging tumor evaluation will be performed every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Women or men aged ≥18 years
3. Histologically or cytologically confirmed adenocarcinoma of the breast with metastatic disease
4. Hormone receptor-negative (ER and PgR < 10%) and HER2-negative (IHC 0,1+ or 2+ ISH not amplified) breast cancer, based on the status of the primary tumor and/or the biopsy of metastatic disease before starting first-line therapy and assessed by local laboratory.
5. Patients ER and PgR < 1% eligible to receive atezolizumab in combination with nab-paclitaxel as standard of care treatment for metastatic triple-negative breast cancer (TNBC), regardless of study participation.
6. PD-L1 positive defined as expression on tumor-infiltrating immune cells ≥1% (SP142 PD-L1 immunohistochemical assay, Ventana Medical Systems), based on the status of the primary tumor and/or the biopsy of metastatic disease before starting first-line therapy and assessed by local laboratory
7. Availability of a representative tumor specimen for translational research
8. Eligible for first-line taxane and carboplatin chemotherapy
9. No prior chemotherapy or targeted systemic therapy (including endocrine therapy) for inoperable locally advanced or metastatic TNBC. Prior radiation therapy for metastatic disease is permitted. There is no required minimum washout period for radiation therapy; however, patients should have recovered from the effects of radiation before enrollment
10. Previous chemotherapy with taxanes and/or carboplatin for early breast cancer (neoadjuvant or adjuvant setting) is permitted if completed ≥12 months before study entry
11. Previous therapy with immune checkpoint inhibitors for early breast cancer (neoadjuvant or adjuvant setting) is permitted if completed ≥12 months before study entry
12. ECOG performance status of 0 or 1
13. Life expectancy ≥ 12 weeks
14. Measurable or evaluable disease as defined by RECIST v1.1.
15. Adequate hematologic and end-organ function, defined by laboratory results obtained within 2 weeks prior to the first study treatment (Cycle 1, Day 1)
16. Negative human immunodeficiency virus (HIV) test at screening
17. Negative hepatitis B surface antigen (HBsAg) test at screening
18. Negative total hepatitis B core antibody (HBcAb) test at screening, or positive HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. The HBV DNA test will be performed only for patients who have a positive HBcAb test
19. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test
20. Women of child bearing potential must agree to either use a contraceptive method with a failure rate of ≤ 1% per year or to remain abstinent (refrain from heterosexual intercourse) during the treatment period and for at least 5 months after the last dose of atezolizumab, or for at least 6 months after the last dose of paclitaxel. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of ≤ 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception
21. Women of child bearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study drug
22. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm

Exclusion Criteria:

1. Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for at least 2 weeks prior to enrollment.
2. Known central nervous system (CNS) disease, except for treated asymptomatic CNS metastases, provided all of the following criteria are met:

   1. No ongoing requirement for corticosteroids as therapy for CNS disease (anticonvulsants at a stable dose are allowed)
   2. No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to enrollment
   3. No evidence of progression or hemorrhage after completion of CNS directed therapy Note: Patients with new asymptomatic CNS metastases detected at the screening scan must receive radiation therapy and/or surgery for CNS metastases. Following treatment, these patients may then be eligible, if all other criteria above are met.
3. Uncontrolled pleural effusion, pericardial effusion, or ascites (Note: patients with indwelling catheters, such as PleurX® are allowed)
4. Uncontrolled tumor-related pain

   1. Patients requiring narcotic pain medication must be on a stable regimen at study entry.
   2. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
   3. Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not presently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
5. Uncontrolled hypercalcemia (>1.5 mmol/L [>6 mg/dL] ionized calcium or serum calcium [uncorrected for albumin] >3 mmol/L [>12 mg/dL] or corrected serum calcium >ULN) or clinically significant (symptomatic) hypercalcemia

   a) Patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history of clinically significant (symptomatic) hypercalcemia are eligible.
6. Malignancies other than TNBC within 5 years prior to enrollment, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer)
7. Pregnant or lactating women, or intending to become pregnant during the study
8. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome)
9. Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within 3 months prior to first dose, unstable arrhythmias, or unstable angina

   1. Patients with a known left ventricular ejection fraction (LVEF) < 40% will be excluded
   2. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
10. Presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third degree heart block, evidence of prior myocardial infarction, or QT interval corrected using Fridericia's formula (QTcF) >470 ms demonstrated by at least two consecutive ECGs
11. Serious infection requiring antibiotics within 2 weeks prior to enrollment, including but not limited to infections requiring hospitalisation or IV antibiotics, such as bacteremia, or severe pneumonia
12. Major surgical procedure within 4 weeks prior to enrollment or anticipation of the need for a major surgical procedure during the study other than for diagnosis Note: Placement of central venous access catheter(s) (e.g., port or similar) is not considered a major surgical procedure and is therefore permitted
13. Treatment with investigational therapy within 30 days prior to initiation of study treatment
14. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
15. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary (CHO) cells or any component of the atezolizumab formulation
16. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis (MS), vasculitis, or glomerulonephritis (Note: Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone and patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible for this study)
17. Prior allogeneic stem cell or solid organ transplantation
18. History of idiopathic pulmonary fibrosis (IPF, including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan. (Note: History of radiation pneumonitis in the radiation field [fibrosis] is permitted)
19. Positive test for human immunodeficiency virus (HIV)
20. Active hepatitis B (positive hepatitis B surface antigen [HBsAg] test or hepatitis B virus [HBV] DNA polymerase chain reaction [PCR] test at screening) or hepatitis C (positive hepatitis C virus antibody test at screening). Note:

    * Patients with past HBV infection or resolved HBV infection (defined as having negative HBsAg and HBV DNA test but a positive hepatitis B core antibody [HBcAb] test) are eligible
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV ribonucleic acid (RNA)
21. Current treatment with anti-viral therapy for HBV
22. Active tuberculosis
23. Receipt of a live, attenuated vaccine within 4 weeks prior to enrollment or anticipation that such a live, attenuated vaccine will be required during the study Note: Patients must agree not to receive live, attenuated influenza vaccine (e.g., FluMist®) within 28 days prior to enrollment, during treatment or within 5 months following the last dose of atezolizumab
24. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug (whichever is longer) prior to enrollment
25. Treatment with systemic immunosuppressive medications (including but not limited to corticosteroids, cyclophosphamide, azathioprine, cyclosporine, methotrexate, thalidomide, and antitumour necrosis factor [TNF] agents) within 2 weeks prior to enrollment, or anticipated requirement for systemic immunosuppressive medications during the trial

    1. Patients who have received acute, low-dose (≤ 10 mg oral prednisone or equivalent), systemic immunosuppressant medications may be enrolled in the study
    2. Patients with a history of allergic reaction to IV contrast requiring steroid pretreatment should have baseline and subsequent tumor assessments performed using MRI
    3. The use of corticosteroids (≤ 10 mg oral prednisone or equivalent) for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low dose supplemental corticosteroids for adrenocortical insufficiency are allowed
26. Poor peripheral venous access
27. Illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
28. Any other serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
29. History of hypersensitivity reactions to paclitaxel or other drugs formulated in the same solvent as nab-paclitaxel
30. History of hypersensitivity reactions to carboplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2024-07-03 (Estimated); Study Completion 2024-07-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  % Overall survival

SECONDARY OUTCOMES:
Overall survival | 2,5 years
  % Overall survival
Overall survival in HR | 2 years
  OS in HR <1% and in HR 1-10%
Post-progression survival | up 24 months from LPFV (from tumor progression until death or is censored on the date of the last follow-up consultation up to 24 months)
  obrservation of Post-progression survival
Objective response rate | from 12 weeks to 24 months (An objective response is defined for patients with measurable disease at baseline as either a partial response (PR) or a complete response (CR) using RECIST v1.1 up to 24 months)
  observation of Objective response rate
Time to treatment failure | from 4 weeks to 24 months (Time to treatment failure (TTF) is defined as the time from enrollment to treatment discontinuation for any reason, including disease progression, treatment toxicity, patient preference, or death up to 24 months)
  observation of Time to treatment failure
Incidence and severity od AEs and SAEs | up to 24 months
  Incidence and severity of adverse events and serious adverse events

OTHER OUTCOMES:
Exploratory outcome | continuosly during the study up to 24 months from LPFV
  Variation of ctDNA levels from baseline to first evaluation through the multigene FoundationOne® Liquid NGS panel

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Del Mastro, MD, Study Director — San Martino Hospital, Genova
Locations (15):
- Italy (15):
  - Centro di Riferimento oncologico, Aviano, Pordenone
  - A.O. Ospedale Papa Giovanni XXIII - Oncologia, Bergamo
  - Policlinico S. Orsola Malpighi - Oncologia Medica, Bologna
  - Azienda Ospedaliera S. Croce e Carle - Oncologia, Cuneo
  - Arcispedaliera S. Anna di Ferrara U.O. Oncologia Clinica, Ferrara
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - Oncologia ed ematologia clinica e sperimentale, Meldola
  - Istituto Nazionale dei Tumori - Fondazione G. Pascale U.O. Oncologia Medica Senologica, Napoli
  - Università di Napoli Federico II - Facoltà di Medicina Dipartimento di Medicina Clinica e Chirurgia - Oncologia, Napoli
  - Azienda Ospedaliera Universitaria di Parma - Oncologia Medica, Parma
  - IRCCS Arcispedale Santa Maria Nuova - Oncologia Medica, Reggio Emilia
  - Istituto Nazionale Tumori Regina Elena - Oncologia Medica 1, Roma
  - AZIENDA OSPEDALIERA SANTA MARIA TERNI - Oncologia Medica, Terni
  - Presidio San Lazzaro - A.O.U. San Giovanni Battista di Torino (Molinette) - Oncologia, Torino
  - Ospedale Mauriziano Umberto I - Oncologia, Torino
  - ULSS 8 Berica- Ospedale San Bortolo di Vicenza - Oncologia, Vicenza

DOCUMENTS (1):
  • Study Protocol (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT05266937/Prot_000.pdf